CLINICAL TRIAL: NCT03404674
Title: A Phase 1 Dose Escalating Study of a Prototype CS6 Subunit Vaccine With a Modified Heat-labile Enterotoxin From Enterotoxigenic Escherichia Coli (ETEC)
Brief Title: Dose Escalating Study of a Prototype CS6 Subunit Vaccine With a Modified Heat-labile Enterotoxin From Enterotoxigenic Escherichia Coli (ETEC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VAC-050
Record Dates: First submitted 2018-01-10; First posted 2018-01-19 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-11

CONDITIONS: Diarrhea
Keywords: ETEC; Escherichia coli; enteric
MeSH Terms: conditions — Diarrhea; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group A1: CssBA 5 ug (Experimental): Participants received an intramuscular injection of 5 ug CssBA on days 1, 22, and 43.
  Interventions: Biological: CssBA
- Group A2: DmLT 100 ng (Experimental): Participants received an intramuscular injection of 100 ng DmLT on days 1, 22, and 43.
  Interventions: Biological: dmLT
- Group B: CssBA 5 ug + DmLT 100 ng (Experimental): Participants received an intramuscular injection of 5 ug CssBA + 100 ng dmLT on days 1, 22, and 43.
  Interventions: Biological: CssBA; Biological: dmLT
- Group C: CssBA 5 ug + DmLT 500 ng (Experimental): Participants received an intramuscular injection of 5 ug CssBA + 500 ng dmLT on days 1, 22, and 43.
  Interventions: Biological: CssBA; Biological: dmLT
- Group D: CssBA 15 ug + DmLT 500 ng (Experimental): Participants received an intramuscular injection of 15 ug CssBA + 500 ng dmLT on days 1, 22, and 43.
  Interventions: Biological: CssBA; Biological: dmLT
- Group E: CssBA 45 ug + DmLT 500 ng (Experimental): Participants received an intramuscular injection of 45 ug CssBA + 500 ng dmLT on days 1, 22, and 43.
  Interventions: Biological: CssBA; Biological: dmLT

INTERVENTIONS:
Biological: CssBA — Recombinant enterotoxigenic Escherichia coli (ETEC) surface antigen 6 containing modified structural subunits A and B
  Other Names: spd_dsc16Bntd14CssBAB7A[His]₆
  Arms: Group A1: CssBA 5 ug; Group B: CssBA 5 ug + DmLT 100 ng; Group C: CssBA 5 ug + DmLT 500 ng; Group D: CssBA 15 ug + DmLT 500 ng; Group E: CssBA 45 ug + DmLT 500 ng
Biological: dmLT — Escherichia coli double mutant heat-labile toxin with mutations at amino acids 192 and 211
  Arms: Group A2: DmLT 100 ng; Group B: CssBA 5 ug + DmLT 100 ng; Group C: CssBA 5 ug + DmLT 500 ng; Group D: CssBA 15 ug + DmLT 500 ng; Group E: CssBA 45 ug + DmLT 500 ng

SUMMARY:
This study will evaluate the safety of a prototype Coli surface antigen 6 (CS6) subunit vaccine (CssBA) alone or in combination with Escherichia coli double mutant heat labile toxin (dmLT) given by intramuscular (IM) injection.

DETAILED DESCRIPTION:
This is an open-label clinical trial in which a total of 50 participants will receive three injections of either CssBA alone, dmLT alone or CssBA + dmLT. The vaccine will be administered via IM injection to alternating deltoid regions on days 1, 22, and 43. Each participant will receive the same dose at each vaccination dependent upon group assignment. Group A is considered a pilot group in which all 3 doses will be administered and participants monitored for safety 7 days after the third vaccination, prior to the enrollment of participants in Group B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
2. Completion and review of comprehension test (achieved > 70% accuracy).
3. Signed informed consent document.
4. Available for the required follow-up period and scheduled clinic visits.
5. Women: Negative pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within three (3) months following last vaccination.

Exclusion Criteria:

1. Health problems (for example, intercurrent febrile illness, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension or any other condition that might place the subject at increased risk of adverse events) - study clinicians, in consultation with the PI, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the Research Monitor as appropriate.
2. Clinically significant abnormalities on physical examination.
3. Immunosuppressive drugs (use of systemic corticosteroids or chemotherapeutics that may influence antibody development) or illness (including immunoglobulin A [IgA] deficiency, defined by serum IgA < 7 mg/dL).
4. Women who are pregnant or planning to become pregnant during the study period plus three (3) months beyond the last received dose and currently nursing women.
5. Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) 30 days before planned date of first vaccination or anytime through the last study safety visit.
6. Positive blood test for Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV), human immunodeficiency virus (HIV)-1/2.
7. Clinically significant abnormalities on basic laboratory screening.
8. Exclusionary skin disease history/findings that would confound assessment or prevent appropriate local monitoring of adverse events (AEs), or possibly increase the risk of a local AE
9. History of chronic skin disease (clinician judgement)
10. Acute skin infection/eruptions on the upper arms including fungal infections, severe acne or active contact dermatitis
11. Allergies that may increase the risk of AEs
12. Regular use (weekly or more often) of antidiarrheal, anti-constipation, or antacid therapy
13. Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis
14. History of microbiologically confirmed ETEC or cholera infection in the last 3 years
15. Travel to countries where ETEC or V. cholerae or other enteric infections are endemic (most of the developing world) within 3 years prior to dosing (clinician judgement)
16. Symptoms consistent with Travelers' Diarrhea or concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study
17. Vaccination for or ingestion of ETEC, cholera, or E. coli heat labile toxin within 3 years prior to dosing
18. Occupation involving handling of ETEC or V. cholerae currently, or in the past 3 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tida K Lee, MD, PhD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research Clinical Trial Center, Silver Spring, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult men and women, civilian and active-duty military, were recruited from the Baltimore/Washington, DC area through the Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center (CTC) by the use of advertisement in multiple media formats.
Pre-assignment Details: Participants were sequentially enrolled to received either recombinant enterotoxigenic Escherichia coli (ETEC) surface antigen 6 vaccine (CssBA) alone, Escherichia coli double mutant heat-labile toxin (dmLT) alone, or CssBA co-administered with dmLT. Participants were to receive 3 vaccinations at the same dose of their assigned treatment.
  Enrollment of subsequent groups was dependent on safety measured in the first 7 days after the third vaccination of the previous group.
Groups:
- Group A1: CssBA 5 µg: Participants received an intramuscular injection of 5 µg CssBA on days 1, 22, and 43.
- Group B: CssBA 5 µg + DmLT 100 ng: Participants received an intramuscular injection of 5 µg CssBA co-administered with 100 ng dmLT on days 1, 22, and 43.
- Group C: CssBA 5 µg + DmLT 500 ng: Participants received an intramuscular injection of 5 µg CssBA co-administered with 500 ng dmLT on days 1, 22, and 43.
- Group D: CssBA 15 µg + DmLT 500 ng: Participants received an intramuscular injection of 15 µg CssBA co-administered with 500 ng dmLT on days 1, 22, and 43.
- Group E: CssBA 45 µg + DmLT 500 ng: Participants received an intramuscular injection of 45 µg CssBA co-administered with 500 ng dmLT on days 1, 22, and 43.
Period: Overall Study
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Started (Enrolled and received Dose 1) | 5 | 5 | 10 | 10 | 10 | 10
Received Dose 2 | 5 | 4 | 10 | 9 | 10 | 10
Received Dose 3 | 5 | 4 | 9 | 9 | 10 | 9
Completed | 5 | 4 | 8 | 9 | 10 | 9
Not Completed | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Inability to Attend Future Visits | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Behavioral Problems | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Started a Medication that Precluded Eligibility | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng | Total
Number analyzed (Participants) | 5 | 5 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [30 to 41] | 29 [27 to 37] | 29.5 [26 to 32] | 31.5 [27 to 37] | 28 [22 to 38] | 29.5 [25 to 33] | 30 [26 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 7 | 5 | 7 | 30
  Male | 1 | 3 | 5 | 3 | 5 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 2 | 1 | 6
  Not Hispanic or Latino | 5 | 3 | 9 | 10 | 8 | 9 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Black | 4 | 4 | 3 | 5 | 3 | 4 | 23
  White | 1 | 1 | 7 | 3 | 7 | 5 | 24
  Multi-race | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10 | 10 | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events
Description: Solicited adverse events included vaccine site pain, vaccine site pruritus, vaccine site rash/eruption, vaccine site swelling, vaccine site tenderness, fever, headache, diarrhea, arthralgia, myalgia, malaise, nausea, and vomiting.
  Adverse events were assessed for severity by the investigator according to the following:
  Mild (Grade 1): Does not interfere with routine activities, minimal level of discomfort
  Moderate (Grade 2): Interferes with routine activities, moderate level of discomfort
  Severe (Grade 3): Unable to perform routine activities, significant level of discomfort
  Potentially life-threatening (Grade 4): Hospitalization or emergency room (ER) visit for potentially life-threatening event
Time Frame: From first vaccination to 28 days after the third vaccination, 71 days.
Population: All participants who received one or more doses of the study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 5 | 10 | 10 | 10 | 10
Participants
  Mild | 2 | 5 | 9 | 9 | 10 | 10
  Moderate | 0 | 0 | 2 | 1 | 2 | 2
  Severe | 0 | 0 | 0 | 0 | 1 | 0
  Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With a Serum Immunologic Response to Coli Surface Antigen 6 (CS6)
Description: Serum samples were assayed for immunoglobulin G (IgG) and immunoglobulin A (IgA) antibody titers against CS6 using an enzyme-linked Immunosorbent assay (ELISA). Immunologic response was defined as a ≥ 4-fold increase in reciprocal endpoint titer between Baseline and any post-vaccination sample.
Time Frame: Baseline (Day 1 predose), Days 22 and 43 predose, and Day 70
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available.
Measure: Number; unit: percentage of participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
percentage of participants
  IgA response | 0.0 | 0.0 | 0.0 | 44.4 | 30.0 | 50.0
  IgG response | 20.0 | 0.0 | 77.8 | 100.0 | 100.0 | 90.0

3. Secondary Outcome: Percentage of Participants With a Serum Immunologic Response to Labile Toxin
Description: Serum samples were assayed for immunoglobulin G (IgG) and immunoglobulin A (IgA) antibody titers against labile toxin using an enzyme-linked Immunosorbent assay (ELISA). Immunologic response was defined as a ≥ 4-fold increase in reciprocal endpoint titer between Baseline and any post-vaccination sample.
Time Frame: Baseline (Day 1 predose), Days 22 and 43 predose, and Day 70
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available.
Measure: Number; unit: percentage of participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
percentage of participants
  IgA response | 0.0 | 50.0 | 22.2 | 77.8 | 50.0 | 70.0
  IgG response | 0.0 | 100.0 | 66.7 | 100.0 | 90.0 | 100.0

4. Secondary Outcome: Percentage of Participants With a Mucosal Immunologic Response to Coli Surface Antigen 6 (CS6)
Description: Peripheral blood mononuclear cells (PBMCs) were collected to determine antibody responses from lymphocyte supernatant against CS6 at Baseline and 7 days after each vaccination. Antibody in lymphocyte supernatant (ALS) is an indirect quantification of antibody secreting cells (ASC) activated in the mucosa that circulate in the peripheral blood about seven days post-mucosal immunization/infection. After incubation, lymphocyte supernatant was assayed for antigen-specific IgG and IgA antibodies using ELISA.
  A positive ALS response was defined as a four-fold rise in antibody titers between Baseline and any post vaccination sample.
Time Frame: Baseline (Day 1 pre-dose), Days 8 and 29 predose, and Day 50
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available.
Measure: Number; unit: percentage of participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
percentage of participants
  IgA response | 0.0 | 0.0 | 33.3 | 88.9 | 80.0 | 100.0
  IgG response: number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  IgG response | 60.0 | 0.0 | 100.0 | 88.9 | 100.0 | 80.0

5. Secondary Outcome: Percentage of Participants With a Mucosal Immunologic Response to Labile Toxin
Description: Peripheral blood mononuclear cells (PBMCs) were collected to determine antibody responses from lymphocyte supernatant against labile toxin at Baseline and 7 days after each vaccination. Antibody in lymphocyte supernatant (ALS) is an indirect quantification of antibody secreting cells (ASC) activated in the mucosa that circulate in the peripheral blood about seven days post-mucosal immunization/infection. After incubation, lymphocyte supernatant was assayed for antigen-specific IgG and IgA antibodies using ELISA.
  A positive ALS response was defined as a four-fold rise in antibody titers between Baseline and any post vaccination sample.
Time Frame: Baseline (Day 1 pre-dose), Days 8 and 29 predose, and Day 50
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available.
Measure: Number; unit: percentage of participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
percentage of participants
  IgA response | 0.0 | 100.0 | 22.2 | 77.8 | 90.0 | 100.0
  IgG response: number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  IgG response | 0.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

6. Secondary Outcome: Geometric Mean Titer of Serum Anti-CS6 Immunoglobulin G Antibodies
Description: Serum samples were assayed for IgG antibody titers against CS6 using an enzyme-linked Immunosorbent assay (ELISA).
Time Frame: Days 1, 22, and 43 pre-vaccination, and Day 70
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available, and with available data at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 39.0 [18.2 to 83.6] | 29.6 [17.5 to 50.1] | 39.1 [22.2 to 69.1] | 36.9 [20.5 to 66.6] | 40.5 [24.6 to 66.7] | 51.5 [26.1 to 101.4]
  Day 22 (pre-vaccination) | 40.2 [17.8 to 90.8] | 34.1 [12.9 to 90.7] | 28.2 [21.6 to 36.8] | 81.2 [16.6 to 396.6] | 80.1 [39.4 to 162.9] | 107.1 [28.3 to 405.7]
  Day 43 (pre-vacination) | 57.4 [16.9 to 195] | 46.6 [14.5 to 149.8] | 108.9 [54.3 to 218.4] | 513.5 [77.2 to 3415.4] | 288.2 [100.2 to 829.2] | 958.3 [235.9 to 3893.4]
  Day 70 (28 days after last vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 70 (28 days after last vaccination) | 81.3 [19.0 to 346.7] | 29.4 [17.8 to 48.5] | 695.3 [182.1 to 2655.3] | 4631.2 [1462.3 to 14667.6] | 2520.4 [1199.2 to 5297.2] | 5167.1 [1298.8 to 20556.8]

7. Secondary Outcome: Geometric Mean Titer of Serum Anti-CS6 Immunoglobulin A Antibodies
Description: Serum samples were assayed for IgA antibody titers against CS6 using an enzyme-linked Immunosorbent assay (ELISA).
Time Frame: Days 1, 22, and 43 pre-vaccination, and Day 70
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 269.9 [133.6 to 545.1] | 213.4 [73.0 to 623.6] | 308.5 [181.4 to 524.4] | 330.0 [176.1 to 618.6] | 368.2 [192.3 to 705.0] | 370.8 [180.9 to 760.0]
  Day 22 (pre-vaccination) | 294.3 [128.7 to 672.9] | 215 [64.9 to 712.4] | 285.1 [172.9 to 469.9] | 846.9 [189.1 to 3792.6] | 408.0 [223.1 to 746.1] | 523.5 [262.0 to 1045.9]
  Day 43 (pre-vacination) | 260.9 [122.0 to 557.8] | 164.7 [47.5 to 571.3] | 328.7 [200.5 to 538.8] | 1571.0 [341.7 to 7222.1] | 505.2 [275.8 to 925.4] | 1188.9 [515.4 to 2742.6]
  Day 70 (28 days after last vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 70 (28 days after last vaccination) | 339.1 [143.6 to 800.6] | 218.0 [48.4 to 982.4] | 521.6 [236.5 to 1150.3] | 2483.1 [595.3 to 10357.2] | 970.3 [553.4 to 1701.4] | 2170.4 [1053.0 to 4473.7]

8. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Adverse events were assessed for severity by the investigator according to the following:
  Mild (Grade 1): Does not interfere with routine activities Minimal level of discomfort
  Moderate (Grade 2): Interferes with routine activities Moderate level of discomfort
  Severe (Grade 3): Unable to perform routine activities Significant level of discomfort
  Potentially life-threatening (Grade 4): Hospitalization or emergency room (ER) visit for potentially life-threatening event
Time Frame: From first vaccination to 28 days after the third vaccination, 71 days.
Population: All participants who received one or more doses of the study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 5 | 10 | 10 | 10 | 10
Participants
  Mild | 4 | 3 | 5 | 6 | 10 | 9
  Moderate | 2 | 0 | 2 | 0 | 1 | 3
  Severe | 1 | 0 | 1 | 0 | 1 | 2
  Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Geometric Mean Titer of Serum Anti-LT Immunoglobulin G Antibodies
Description: Serum samples were assayed for IgG antibody titers against labile toxin using an enzyme-linked Immunosorbent assay (ELISA).
Time Frame: Days 1, 22, and 43 pre-vaccination, and Day 70
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 46.1 [16.4 to 129.7] | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 84.5 [31.8 to 224.0] | 88.9 [54.0 to 146.5] | 75.0 [37.4 to 150.4] | 48.8 [25.0 to 95.2]
  Day 22 (pre-vaccination) | 48.3 [15.3 to 152.1] | 52.8 [11.4 to 243.9] | 172.9 [42.4 to 705.5] | 1010.3 [182.9 to 5579.8] | 235.0 [64.1 to 860.7] | 193.2 [80.0 to 466.6]
  Day 43 (pre-vacination) | 46.3 [15.8 to 136.0] | 303.7 [39.8 to 2316.2] | 235.6 [67.5 to 822.0] | 2671.0 [754.2 to 9459.1] | 679.2 [256.7 to 1797.0] | 666.8 [339.7 to 1308.9]
  Day 70 (28 days after last vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 70 (28 days after last vaccination) | 55.0 [17.8 to 170.1] | 398.1 [91.9 to 1724.3] | 424.1 [159.7 to 1126.6] | 3114.1 [965.3 to 10046.6] | 1116.9 [467.8 to 2666.7] | 1086.4 [473.8 to 2491.2]

10. Secondary Outcome: Geometric Mean Titer of Serum Anti-LT Immunoglobulin A Antibodies
Description: Serum samples were assayed for IgA antibody titers against labile toxin using an enzyme-linked Immunosorbent assay (ELISA).
Time Frame: Days 1, 22, and 43 pre-vaccination, and Day 70
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 28.4 [21.4 to 37.7] | 25.8 [24.2 to 27.6] | 28.6 [21.3 to 38.5] | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero
  Day 22 (pre-vaccination) | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 30.4 [16.6 to 55.6] | 55.8 [24.6 to 126.5] | 258.4 [49.3 to 1352.9] | 77.8 [35.3 to 171.3] | 134.6 [57.0 to 317.6]
  Day 43 (pre-vacination) | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 46.2 [9.0 to 238.30] | 48.5 [22.0 to 107.0] | 317.9 [72.8 to 1388.5] | 75.9 [33.6 to 171.4] | 159.6 [62.8 to 405.3]
  Day 70 (28 days after last vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 70 (28 days after last vaccination) | 25.1 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 66.1 [10.6 to 410.1] | 51.4 [20.9 to 126.4] | 202.1 [43.8 to 932.2] | 68.2 [29.9 to 155.6] | 121.1 [57.2 to 256.1]

11. Secondary Outcome: Geometric Mean Titer of Antibody Lymphocyte Supernatant Anti-CS6 Immunoglobulin G Antibodies
Description: Lymphocyte supernatant was assayed for IgG antibody titers against CS6 using ELISA.
Time Frame: Days 1, 8, 29 and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 5.7 [2.5 to 12.8] | 4. [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero
  Day 8 (7 days after 1st vaccination) | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 5.0 [2.9 to 8.6] | 14.9 [3.2 to 70.3] | 8.5 [2.7 to 26.6] | 7.1 [3.0 to 17.0]
  Day 29 (7 days after 2nd vacination) | 6.0 [2.0 to 18.4] | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 42.9 [10.7 to 172.0] | 29.8 [8.2 to 108.6] | 47.4 [12.7 to 176.5]
  Day 50 (7 days after 3rd vaccination) | 18.1 [3.1 to 106.4] | 4.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 86.7 [43.1 to 174.4] | 356.9 [208.5 to 610.7] | 238.3 [115.3 to 492.3] | 142.8 [32.2 to 633.2]

12. Secondary Outcome: Geometric Mean Titer of Antibody Lymphocyte Supernatant Anti-CS6 Immunoglobulin A Antibodies
Description: Lymphocyte supernatant was assayed for IgA antibody titers against CS6 using ELISA.
Time Frame: Days 1, 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [2.5 to 2.5]
  Day 8 (7 days after 1st vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 7.3 [1.3 to 42.2] | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 4.5 [1.9 to 10.8]
  Day 29 (7 days after 2nd vacination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 17.5 [4.0 to 76.0] | 3.3 [1.8 to 6.0] | 33.1 [14.7 to 74.3]
  Day 50 (7 days after 3rd vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 50 (7 days after 3rd vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 6.4 [2.1 to 19.6] | 46.6 [13.8 to 157.2] | 24.1 [8.5 to 68.7] | 35.2 [17.4 to 71.0]

13. Secondary Outcome: Geometric Mean Titer of Antibody Lymphocyte Supernatant Anti-LT Immunoglobulin G Antibodies
Description: Lymphocyte supernatant was assayed for IgG antibody titers against labile toxin using ELISA.
Time Frame: Days 1, 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Group A2: DmLT 100 ng: Participants received 3 intramuscular injections of 100 ng DmLT on days 1, 22, and 43.
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 3.5 [1.6 to 7.8] | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 3.1 [2.0 to 4.8] | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero
  Day 8 (7 days after 1st vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 6.6 [1.5 to 29.2] | 24.0 [6.0 to 97.0] | 47.4 [8.7 to 258.8] | 17.6 [5.0 to 61.4]
  Day 29 (7 days after 2nd vacination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 13.4 [0.6 to 305.9] | 10.0 [2.0 to 49.9] | 105.8 [60.7 to 184.3] | 80.7 [50.2 to 129.9] | 253.5 [116.5 to 551.8]
  Day 50 (7 days after 3rd vaccination) | 2.5 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 88.1 [48.2 to 161.0] | 70.0 [41.5 to 117.9] | 138.4 [102.0 to 187.7] | 123.3 [100.0 to 152.0] | 187.5 [101.9 to 345.0]

14. Secondary Outcome: Geometric Mean Titer of Antibody Lymphocyte Supernatant Anti-LT Immunoglobulin A Antibodies
Description: Lymphocyte supernatant was assayed for IgA antibody titers against labile toxin using ELISA.
Time Frame: Days 1, 8, 29, and 50
Population: Participants who received at least 2 vaccine doses and had at least 2 post-vaccine samples available, and with available samples at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
Number analyzed (Participants) | 5 | 4 | 9 | 9 | 10 | 10
titer
  Day 1 (pre-vaccination) | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.8 [1.3 to 5.9] | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero
  Day 8 (7 days after 1st vaccination) | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 3.0 [1.1 to 8.1] | 11.7 [2.9 to 46.9] | 12.7 [3.8 to 42.8] | 9.0 [2.8 to 28.2]
  Day 29 (7 days after 2nd vacination) | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 9.9 [0.5 to 198.1] | 4.1 [1.4 to 12.4] | 28.7 [8.8 to 93.9] | 19.3 [7.9 to 47.3] | 60.5 [44.9 to 81.6]
  Day 50 (7 days after 3rd vaccination): number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 10
  Day 50 (7 days after 3rd vaccination) | 2.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 13.3 [1.6 to 107.6] | 3.6 [1.4 to 9.5] | 24.7 [7.6 to 80.0] | 23.6 [8.5 to 65.4] | 18.7 [5.8 to 60.5]

ADVERSE EVENTS:
Time Frame: From the day of the first vaccination up to 28 days after the third vaccination, 71 days.
Arm/Group | Group A1: CssBA 5 µg | Group A2: DmLT 100 ng | Group B: CssBA 5 µg + DmLT 100 ng | Group C: CssBA 5 µg + DmLT 500 ng | Group D: CssBA 15 µg + DmLT 500 ng | Group E: CssBA 45 µg + DmLT 500 ng
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5 | 10/10 | 10/10 | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A1: CssBA 5 µg (N=5) | Group A2: DmLT 100 ng (N=5) | Group B: CssBA 5 µg + DmLT 100 ng (N=10) | Group C: CssBA 5 µg + DmLT 500 ng (N=10) | Group D: CssBA 15 µg + DmLT 500 ng (N=10) | Group E: CssBA 45 µg + DmLT 500 ng (N=10)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 1
Conjunctivital hemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hemorroidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Axillary Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hangover (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaccination Site Bruising (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Vessel Puncture Site Hematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vessel Puncture Site Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1 | 1 | 2 | 6
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0
Hemoglobin decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 2
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diastolic Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Systolic Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 3 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 3 | 0 | 3 | 2
Pyrexia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vaccination Site Pain (General disorders) | 0 | 1 | 2 | 5 | 9 | 9
Vaccination Site Pruritus (General disorders) | 0 | 0 | 1 | 1 | 7 | 0
Vaccination Site Discoloration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination Site Erythema (General disorders) | 1 | 4 | 7 | 7 | 8 | 8
Vaccination Site Induration (General disorders) | 0 | 0 | 0 | 6 | 5 | 6
Vaccination Site Papule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination Site Swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 4
Headache (Nervous system disorders) | 1 | 0 | 6 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT03404674/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03404674/SAP_001.pdf